CLINICAL TRIAL: NCT02123732
Title: Role of DbXell in the Treatment of Subjects With Mildly Uncontrolled Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laniado Hospital (Other)
Collaborators: KGS Research (Other)
Responsible Party: Principal Investigator, Laniado Hospital, Dr Mark J NIVEN Director of Endocrine and Diabetes Unit, Laniado Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DbXell1234
Record Dates: First submitted 2014-04-02; First posted 2014-04-28 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Diabetes Mellitus; Herbal; food supplement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DbXell (Experimental): Drug: DbXell three times daily for 12 weeks and then switching to Placebo of DbXell for 12 additional months Other: Lifestyle modification Each study subject will be provided with and instructed to follow a lifestyle modification (particularly regarding dietary advice and exercise) during the subject's participation in the study.
  Interventions: Dietary Supplement: DbXell
- Placebo (Placebo Comparator): Drug: Placebo of DbXell Placebo of DbXell three times daily for 12 weeks and then switching to DbXell for 12 additional weeks Other: Lifestyle modification Each study subject will be provided with and instructed to follow a lifestyle modification (particularly regarding dietary advice and exercise) during the subject's participation in the study.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DbXell
  Arms: DbXell
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This is a 2-arm, single-blind, crossover, placebo-controlled clinical study, with 24 weeks of therapy to evaluate the efficacy and safety of DbXell in improving metabolic control in patients with Type 2 Diabetes that is mildly uncontrolled, defined as HbA1c above target but less than 8.0% on their current conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age of 18-70 years Established type 2 diabetes mellitus as defined by the American Diabetes Association, but of duration less than 10 years.
* Suboptimal glycemic control as judged by HbA1c over target but not more than 8.0%.Current medication of not more than 2 oral hypoglycemic agents. No current or past insulin or GLP1 therapy.
* FPG ≤ 180 mg/dL
* Hemoglobin level of ≥ 10.0 g/dL
* Serum ALT ≤ 2.5 times upper limit of normal
* Serum creatinine < 1.5 times upper limit of normal

Exclusion Criteria:

* Female of childbearing potential
* Subjects with symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other symptomatic ischemic arterial diseases necessitating medical treatment
* Uncontrolled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg)
* History of renal and/or liver disease
* History of or the presence of any clinical evidence of malignancies
* Presence of exacerbation of chronic illnesses, severe and acute infections, complicated infections
* Current treatment with systemic corticosteroids or herbal (alternative) medicines
* Participation in any other intervention trial within 30 days prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C concentrations and fasting glucose levels | 6 months from last patient in

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Niven, MD, Principal Investigator — Laniado Hospital
Locations (1):
- Laniado Hospital, Diabetes Unit, Netanya, Israel